CLINICAL TRIAL: NCT00566475
Title: School Centered Telemedicine Program for Children With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); New York State Department of Health (Other Government); Children's Miracle Network (Other)
Responsible Party: Principal Investigator, Roberto Izquierdo, Professor of Medicine and Pediatrics, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#5302
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2017-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Usual care of type 1 diabetes at the diabetes center
- 2 (Experimental): Usual care at the diabetes center supplemented by a telemedicine intervention in the school involving school personnel, the child with diabetes and at least 1 parent of the child. The diabetes center NP conducts videovisits with the school nurse, patient (child) +/- parent monthly.
  Interventions: Other: telemedicine

INTERVENTIONS:
Other: telemedicine — School telemedicine intervention involving school personnel, the child with type 1 diabetes and at least 1 parent
  Arms: 2

SUMMARY:
The purpose of this study is to determine if using school-based telemedicine for diabetes support and education in students with type 1 diabetes in grades K-8 can lead to improvement in control of diabetes and improved satisfaction of all caregivers.

DETAILED DESCRIPTION:
Subjects, ages 5 to 14 years (grades kindergarten through eighth) were randomized to usual care (18 students; 13 schools) or intervention (23 students; 12 schools). Usual care included medical visits every 3 months and communication between school nurse and diabetes team as needed by phone. The intervention group received usual care plus a telemedicine unit in the school nurse office to videoconference between the school nurse, child, and diabetes team every month. Hemoglobin A1c and pediatric quality of life were measured every 3 months for 1 year. Analyses used multilevel modeling.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes under care of Joslin Diabetes Center in Syracuse NY
* Grade K-8
* Age 5-14 at time of enrollment
* Consent of student, parent and school

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c | 1 year

SECONDARY OUTCOMES:
glucose levels, hypoglycemia, quality of life, satisfaction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ruth S Weinstock, MD PhD, Principal Investigator — State University of New York - Upstate Medical University; Roberto E Izquierdo, MD, Study Director — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Result] Izquierdo R, Morin PC, Bratt K, Moreau Z, Meyer S, Ploutz-Snyder R, Wade M, Weinstock RS. School-centered telemedicine for children with type 1 diabetes mellitus. J Pediatr. 2009 Sep;155(3):374-9. doi: 10.1016/j.jpeds.2009.03.014. Epub 2009 May 21. PMID 19464030